CLINICAL TRIAL: NCT04859023
Title: Comparison of Strategies Based on RT-PCR or Antigenic Test for the Screening of SARS-CoV-2 Infection in General Population Using Self-samples (COVID-19).
Brief Title: Comparison of Strategies Based on RT-PCR or Antigenic Test for the Screening of SARS-CoV-2 Infection (COVID-19).
Acronym: AutoCoV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21CH037; 2021-A00390-41 (Other: ANSM)
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: SARS-CoV Infection
Keywords: Covid19; RT-PCR; rapid antigenic test; SARS-CoV-2; self-sampling; diagnosis; mass screening; isolation measures; health education
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Disease; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mass screening SARS-COV-19 (Experimental): 20 0000 participant will be included during mass screening SARS-COV-19 of the population of the city of Saint-Etienne.
  They will have two strategies both based on self-samples: (i) a saliva sample combined to an anterior nare self-swabbing tested by antigenic test versus (ii) a saliva sample tested by RT-PCR.
  Interventions: Diagnostic Test: saliva sample combined to an anterior nare self-swabbing (Self-samples); Diagnostic Test: saliva sample (Self-sample); Other: Survey of SARS-COV-19 knowledge; Other: Survey of acceptability of the different self-samples.

INTERVENTIONS:
Diagnostic Test: saliva sample combined to an anterior nare self-swabbing (Self-samples) — Tested by antigenic test.
Diagnostic Test: saliva sample (Self-sample) — Tested by RT-PCR.
Other: Survey of SARS-COV-19 knowledge — collection of : socio-professional characteristics, questions on health literacy on the transmission of the virus and barrier gestures, adherence to barrier gestures, isolation modalities in case of positivity, motivations for participating in this screening campaign.
Other: Survey of acceptability of the different self-samples. — collection of : assessment and acceptability of the tolerance of self-samples.

SUMMARY:
The virological diagnosis of SARS-CoV-2 infection is pivotal for the control of the outbreak by large screening of a- or pauci-symptomatic subjects. Despite nasopharyngeal swabbing tested by RT-PCR is considered as the gold standard, new strategies based on self-samples are considered as valuable alternatives because of their non-invasiveness and ability to be performed in the absence healthcare worker, especially when the subject is asymptomatic and needs to be tested repetitively. The aim of the present project is to evaluate two strategies both based on self-samples: (i) a saliva sample combined to an anterior nare self-swabbing tested by antigenic test versus (ii) a saliva sample tested by RT-PCR. The comparison will be performed during a mass screening of the population of the city of Saint-Etienne (170000 inhabitants), France. The sensitivity of the rapid antigenic test will be evaluated in comparison to that of RT-PCR considered as gold standard.

DETAILED DESCRIPTION:
The main objective is to evaluate the performance of a strategy for screening for CoV-2-SARS infection that would combine 1) a salivary self-sample with an anterior nasal swab and 2) a diagnostic antigenic test, in comparison with the reference salivary RT-PCR technique recently validated by National Authority for Health (HAS).

ELIGIBILITY:
Inclusion Criteria:

* Adult age or at least 10 year old able to perform self-sampling of saliva and anterior nare swabbing
* Subject or legal tutor agreeing to participate to self-sampling and to collect anonymized data required by the present research

Exclusion Criteria:

* Inability to understand the protocol (language barrier notably)
* Deny to participate to the proposed research
* Patients under tutorship

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Positivity of self-samples combining saliva and anterior nare specimens tested by rapid antigenic test compared to saliva tested by RT-PCR (gold-standard). | Day: 7
  Measured by antigenic test results and RT-PCR results.

SECONDARY OUTCOMES:
Number and percentage of SARS-CoV-2 infection in the selected population tested by reference RT-PCR on saliva | Day: 7
  Measured by RT-PCR results.
Number and percentage of the circulation of different variants of interest of SARS-CoV-2 viruses in the tested population | Day: 7
  Measured by RT-PCR results.
Evaluate the acceptability (pain, discomfort, speed of execution) of self-samples according to age and socio-professional categories | Day: 7
  Measured by survey of acceptability of the different self-samples results.
Evaluate the cost-effectiveness ratio of the new strategy by comparison to the gold standard (RT-PCR on saliva) | Day: 7
  Measured by number of test performed and performances of self-samples combining saliva and anterior nare specimens tested by rapid antigenic test compared to saliva tested by RT-PCR.
Number of people who have benefited from sensitization and support specifically set up as part of the screening campaign | Day: 7
  Measured the screening day.
Number of persons cared for by the territorial isolation support cell (CTAI) | Day: 7
  Measured the screening day.
Health literacy questionnaire | Day: 7
  It is a questionnaire with items on the transmission of the virus and barrier gestures, adherence to barrier gestures, modalities of isolation in case of positivity and motivations for participating in this screening campaign.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno POZZETTO, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verot E, Bonjean P, Chaux R, Gagnaire J, Gagneux-Brunon A, Pozzetto B, Berthelot P, Botelho-Nevers E, Chauvin F. Development and Validation of the COVID-19 Knowledges and Behavior Questionnaire in a French Population (CoVQuest-CC). Int J Environ Res Public Health. 2022 Feb 23;19(5):2569. doi: 10.3390/ijerph19052569. PMID 35270262